CLINICAL TRIAL: NCT02670577
Title: Measuring the Impact of MammaPrint on Adjuvant and Neoadjuvant Treatment in Breast Cancer Patients: A Prospective Registry
Acronym: IMPACt
Status: Completed | Type: Observational
Sponsor: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: IMPACt
Record Dates: First submitted 2016-01-27; First posted 2016-02-02 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: stage I; stage II; HER2 positive; Triple Negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- stage I or II HR-positive, HER2-negative: Histologically proven invasive stage I and II breast cancer and Hormone Receptor positive & HER2 negative
  & Axillary lymph node status: 0-3 involved
- HER2+: Histologically proven invasive T1a or T1b breast cancer
  & Hormone receptor negative or positive
  & HER2 positive
  & Axillary lymph node status: 0-1 involved
- Triple Negative: Histologically proven invasive T1a or T1b breast cancer
  & Hormone receptor negative
  & HER2 negative
  & Axillary lymph node status: 0-1 involved
- Neoadjuvant: Stage I or II patients receiving neoadjuvant therapy.

SUMMARY:
The scope of this study is to measure the impact of MammaPrint on treatment in Hormone Receptor (HR)-positive HER2-negative breast cancer patients.

In addition, the impact of MammaPrint on treatment in patients with T1a/T1b and pN0/pN1 (up to 1 node), Triple Negative or HER2-positive tumors will be assessed.

DETAILED DESCRIPTION:
Eligible patients will have their tumor sample analyzed for MammaPrint, BluePrint and TargetPrint. Patients cannot start treatment before the MammaPrint and BluePrint result is received and taken into consideration for the treatment plan. The clinical data are to be entered online. There will be 2 Case Report Forms (CRFs). Baseline clinical data and physician chemotherapy intention before knowing the MammaPrint and BluePrint result will be entered in CRF 1. After completion of CRF1, the MammaPrint and BluePrint result will be released. CRF2 will be completed after the final treatment decision has been made. This CRF will capture physician chemotherapy intention after the MammaPrint and BluePrint result and the impact of these results.

A sample size of 331 patients is required to detect a 25% overall treatment change (5% significance and 95% power) in stage I and II HR-positive, HER2-negative patients receiving adjuvant therapy.

In addition at least 50 T1a/bN0/1 (up to 1 node) Triple Negative, at least 50 T1a/bN0/1 (up to 1 node) HER2-positive breast cancer patients, and at least 50 patients receiving neoadjuvant therapy will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive chemotherapy and endocrine therapy as defined by a good Karnofsky index (≥80) and no hematologic, cardiologic or hepatic contraindications, nor any impeding comorbidity
* Informed consent form signed on the same day or before enrollment
* ≥ 18 years of age at time of consent Per study arm
* Histologically proven invasive stage I and II breast cancer and Hormone Receptor positive (ER+ PR-, ER- PR+ or ER+ PR+) according to local standards & HER2 negative: IHC 0-1+, or FISH or other ISH non-amplified (locally assessed)

IMPACt study; version 1 2015 September 1 Page 10 Axillary lymph node status: 0-3 involved (macro metastases i.e. >2mm OR micro metastases i.e. >0.2-2mm)

OR

Histologically proven invasive T1a or T1b breast cancer & Hormone receptor negative (ER- and PR-) according to local standards & HER2 negative: IHC 0-1+, or FISH or other ISH non-amplified (locally assessed)

& Axillary lymph node status: 0-1 involved (macro metastases i.e. >2mm OR micro metastases i.e. >0.2-2mm)

OR

Histologically proven invasive T1a or T1b breast cancer

& Hormone receptor negative or positive (ER-PR-, ER+PR-, ER-PR+, ER+PR+) according to local standards

& HER2 positive: IHC 3+, or FISH or other ISH amplified (locally assessed)

& Axillary lymph node status: 0-1 involved (macro metastases i.e. >2mm OR micro metastases i.e. >0.2-2mm)

Exclusion Criteria:

* Previous diagnosis of breast malignancy unless disease free for 10 years
* Metastatic disease
* Tumor sample shipped to Agendia with ≤ 30% tumor cells or that fails QA or QC criteria
* Women who have started or completed adjuvant chemotherapy or neo-adjuvant chemotherapy for current breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage I or II HR-positive, HER2-negative breast cancer patients AND T1a/b, N0/N1 (up to 1 node) Triple Negative, or HER2-positive breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 481 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-04-30 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Decision | 6 weeks
  Compare treatment decision before and after test results.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Desert Regional Medical Center, Palm Springs, California
  - University of Miami, Miami, Florida
  - St. Joseph's Women's Hospital, Tampa, Florida
  - The Cancer Center at DeKalb Medical, Decatur, Georgia
  - Cadence Cancer Center, Warrenville, Illinois
  - Methodist Hospital, Merrillville, Indiana
  - Community Healthcare System, Munster, Indiana
  - Western Maryland Health System, Cumberland, Maryland
  - Sparrow Cancer Center, Lansing, Michigan
  - Essex Oncology, Belleville, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Akron General Medical Center, Akron, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - St. Clair Hospital, Pittsburgh, Pennsylvania
  - Aurora Cancer Care, Milwaukee, Wisconsin
  - Columbia St. Mary's, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Soliman H, Shah V, Srkalovic G, Mahtani R, Levine E, Mavromatis B, Srinivasiah J, Kassar M, Gabordi R, Qamar R, Untch S, Kling HM, Treece T, Audeh W. MammaPrint guides treatment decisions in breast Cancer: results of the IMPACt trial. BMC Cancer. 2020 Jan 31;20(1):81. doi: 10.1186/s12885-020-6534-z. PMID 32005181